CLINICAL TRIAL: NCT05315505
Title: Effectiveness of a Home-based Pulmonary Rehabilitation Program in COPD Patients
Acronym: Rehab2life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Matosinhos, EPE (Other)
Responsible Party: Principal Investigator, Liliana Silva, RN, Unidade Local de Saúde de Matosinhos, EPE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136/CES/JAS
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation
Keywords: COPD; Pulmonary rehabilitation; Maintenance pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise; Self-Management

STUDY DESIGN:
Intervention Model Description: Randomization will be performed after verifying the inclusion and exclusion criteria in the study and the informed, free and informed consent of the individuals. Randomization will be carried out by permuted blocks of 4 to guarantee the same number of participants in each group.
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluation will be performed by a cardiopulmonary technician that has no information about the patient group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance (Experimental): Participants will undergo an initial home-based pulmonary rehabilitation program for eight weeks.
  At the end of the eight weeks, the participants will be randomly assigned into two groups, one receiving the maintenance pulmonary rehabilitation program and the other receiving the usual care.
  The maintenance arm will receive home visits for supervised physical exercise and progressively alternated with phone calls to motivation and feedback
  Interventions: Other: Maintenance programme
- control (Active Comparator): Participants will undergo an initial home-based pulmonary rehabilitation program for eight weeks.
  At the end of the eight weeks, the participants will be randomly assigned into two groups, one receiving the maintenance pulmonary rehabilitation program and the other receiving the usual care.
  The control group will have access to the usual follow.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Maintenance programme — Continuous educational support, exercise training, behaviour change intervention, and self-management.
  Maintenance home-based pulmonary rehabilitation programme for ten months with alternate supervision
  Other Names: Physical exercise; Behaviour change; Self-management
  Arms: Maintenance
Other: Usual Care — No maintenance programme, and the patient has the usual follow-up and medical appointments
  Arms: control

SUMMARY:
The study aims to develop and test the effectiveness of a new home-based pulmonary rehabilitation program comprising two distinct phases, the first in which an 8-week respiratory rehabilitation program is carried out the second in which a maintenance pulmonary rehabilitation program is carried out.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnose with B or E characterization according to GOLD criteria;
* Residence in the area covered by the institution where the study is carried out

Exclusion Criteria:

* Frequency of a PR programme in the previous six months
* COPD exacerbation for less than one week;
* Presence of unstable comorbidities (List of predetermined diagnoses that constitute absolute exclusion criteria);
* Presence of comorbidities that constitute relative exclusion criteria through a medical evaluation.
* Score of the Clinical Frailty Scale 2.0 above six or above five in case of not having a responsible caregiver and living alone
* SpO2 below 85% in the 6-minute walk test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Distance in meters covered over a time of 6 minutes 0 | Baseline
  Distance in meters covered over a time of 6 minutes 0 measured with the 6 minute walking test (6MWT) - The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Distance in meters covered over a time of 6 minutes 1 | 8 weeks
  Distance in meters covered over a time of 6 minutes 1 measured with the 6 minute walking test (6MWT) - The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Distance in meters covered over a time of 6 minutes 2 | 7 months
  Distance in meters covered over a time of 6 minutes 2 measured with the 6 minute walking test (6MWT) - The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Distance in meters covered over a time of 6 minutes 3 | 12 months
  Distance in meters covered over a time of 6 minutes 3 measured with the 6 minute walking test (6MWT) - The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

SECONDARY OUTCOMES:
Dyspnoea 0 | Baseline
  modified Medical Research Council dyspnoea scale (mMRC) - Range from 1 to 5, The higher the score, the worst the dyspnoea
Dyspnoea 1 | 8 weeks
  modified Medical Research Council dyspnoea scale (mMRC) - Range from 1 to 5, The higher the score, the worst the dyspnoea
Dyspnoea 2 | 7 months
  modified Medical Research Council dyspnoea scale (mMRC) - Range from 1 to 5, The higher the score, the worst the dyspnoea
Dyspnoea 3 | 12 months
  modified Medical Research Council dyspnoea scale (mMRC) - Range from 1 to 5, The higher the score, the worst the dyspnoea
Health-Related Quality of Life 0 | Baseline
  European quality of life-5 dimensions (EQ5D)
Health-Related Quality of Life 1 | 8 weeks
  European quality of life-5 dimensions (EQ5D)
Health-Related Quality of Life 2 | 7 months
  European quality of life-5 dimensions (EQ5D)
Health-Related Quality of Life 3 | 12 months
  European quality of life-5 dimensions (EQ5D)
Number of emergency department visits due to COPD exacerbation 0 | Baseline
  Number of exacerbations (accessing to emergency department)
Number of emergency department visits due to COPD exacerbation 1 | 8 weeks
  Number of exacerbations (accessing to emergency department)
Number of emergency department visits due to COPD exacerbation 2 | 7 months
  Number of exacerbations (accessing to emergency department)
Number of emergency department visits due to COPD exacerbation 3 | 12 months
  Number of exacerbations (accessing to emergency department)
COPD symptom control 0 | Baseline
  COPD Assessment Test - Range from 0 to 40. The higher the score, the worst the clinical control
COPD symptom control 1 | 8 weeks
  COPD Assessment Test - Range from 0 to 40. The higher the score, the worst the clinical control
COPD symptom control 2 | 7 months
  COPD Assessment Test - Range from 0 to 40. The higher the score, the worst the clinical control
COPD symptom control 3 | 12 months
  COPD Assessment Test - Range from 0 to 40. The higher the score, the worst the clinical control
Anxiety and Depression 0 | Baseline
  Hospital Anxiety and Depression Scale (HADS) - HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. HADS scoring was done before and after low-vision consultation to see whether there was a change in the scoring
Anxiety and Depression 1 | 8 weeks
  Hospital Anxiety and Depression Scale (HADS) - HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. HADS scoring was done before and after low-vision consultation to see whether there was a change in the scoring
Anxiety and Depression 2 | 7 months
  Hospital Anxiety and Depression Scale (HADS) - HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. HADS scoring was done before and after low-vision consultation to see whether there was a change in the scoring
Anxiety and Depression 3 | 12 months
  Hospital Anxiety and Depression Scale (HADS) - HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. HADS scoring was done before and after low-vision consultation to see whether there was a change in the scoring
Physical activity 0 | Baseline
  Counting steps per day with the pedometer Yamax EX510
Physical activity 1 | 8 weeks
  Counting steps per day with the pedometer Yamax EX510
Physical activity 2 | 7 months
  Counting steps per day with the pedometer Yamax EX510
Physical activity 3 | 12 months
  Counting steps per day with the pedometer Yamax EX510
Functional capacity 0 | Baseline
  Number of times per minute an individual is able to stand up and sit down on a chair standardised for height
Functional capacity 1 | 8 weeks
  Number of times per minute an individual is able to stand up and sit down on a chair standardised for height
Functional capacity 2 | 7 months
  Number of times per minute an individual is able to stand up and sit down on a chair standardised for height
Functional capacity 3 | 12 months
  Number of times per minute an individual is able to stand up and sit down on a chair standardised for height

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Silva, MSc, Principal Investigator — Matosinhos Local Health Unit
Locations (1):
- Unidade Local de Saúde de Matosinhos, Matosinhos Municipality, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva L, Maricoto T, Mota A, Lemos L, Santos M, Cunha H, Azevedo I, Berger-Estilita J, Costa P, Padilha JM. Effectiveness of a home-based pulmonary rehabilitation maintenance programme: the Rehab2Life study protocol. BMC Nurs. 2024 May 21;23(1):338. doi: 10.1186/s12912-024-01999-6. PMID 38773568